CLINICAL TRIAL: NCT02118779
Title: Observational Prolonged Trial in Myotonic Dystrophy Type 1 to Improve Quality of Life Standards, a Target Identification Collaboration
Brief Title: Observational Prolonged Trial in Myotonic Dystrophy Type 1
Acronym: OPTIMISTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: University of Newcastle Upon-Tyne (Other); Ludwig-Maximilians - University of Munich (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Annet Geerlings, Coordinator Trialoffice Neurology, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/NE/0342; 305697 (Other Grant/Funding Number: EU Seventh Framework Programme); 6836 (Other: Sponsor ref)
Record Dates: First submitted 2014-04-11; First posted 2014-04-21 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Myotonic Dystrophy Type 1
Keywords: Myotonic Dystrophy Type 1; DM1; Physical Exercise; Cognitive Behavioural Therapy; Biomarkers
MeSH Terms: conditions — Myotonic Dystrophy; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioural change intervention (Experimental): Cognitive behavioural therapy (CBT) combined with exercise
  Interventions: Behavioral: Behavioural change intervention
- Standard Patient Management (No Intervention): Standard care like usual (i.e. annual checks with neurologist, checks with cardiologist, if needed physical therapy)

INTERVENTIONS:
Behavioral: Behavioural change intervention — The intervention is cognitive behaviour therapy (CBT). The CBT consists of six different modules. All patients will start with individual goal setting and psycho-education about the role of cognitive-behavioural variables in the disabilities patients' experience. The patient formulates his or her treatment goals in concrete terms and later on in the therapy the goals are realised step by step by the patient. The treatment is tailored to the patient's problems: which of the six modules a patient will receive is dependent on the scores on measures that have been collected at baseline assessment. Based on our previous experience with modular interventions we expect that most patients will receive less than four modules.
  Arms: Behavioural change intervention

SUMMARY:
Myotonic dystrophy type1 (DM1) is a rare, inherited, chronic progressive disease as well as an autosomal dominant multisystemic disorder. It is the most common adult form of muscular dystrophy, with a prevalence of approximately 10 per 100,000 people affected. With 733 million people in Europe, we estimate that 75,000 people are DM1 patients in Europe.

The aim of OPTIMISTIC is to improve clinical practice in the management of patients with this rare disease for which no dedicated treatment is currently available. OPTIMISTIC is a multi-centre, randomised controlled trial designed to compare a two component tailored behavioural change intervention to increase physical activity against standard patient management regimes, with particular attention given to the definition of appropriate outcome measures and new clinical guidelines for DM1 management. The two components of the intervention are 1) cognitive behavioural therapy (CBT) and 2) graded physical activity and we will evaluate the intervention's effectiveness and safety against standard patient management.

Participants will be recruited from myotonic dystrophy clinics and neuromuscular centres in France, Germany, the Netherlands and the UK. A total of 286 male and female patients aged 18 years and older with genetically proven classical or adult DM1 suffering from severe fatigue (only DM1 patients with a CIS subscale fatigue score > 35 are likely to benefit from the intervention), able to walk independently and able to complete the trial interventions will be included.

A key objective of OPTIMISTIC is to provide outcome measures that are relevant for the patients and have a rate of change that is appropriate for a clinical trial timeframe. In addition, OPTIMISTIC will identify genetic factors that predict outcome and potential biomarkers as surrogate outcome measures that best explain the observed clinical variation.

DETAILED DESCRIPTION:
Background DM1 is a rare, inherited, progressive disease as well as an autosomal dominant multisystemic disorder. It is the most common adult form of muscular dystrophy, with a prevalence of approximately 10 per 100,000 people affected. With 733 million people in Europe, we estimate that 75,000 people are DM1 patients in Europe. Typical symptoms of the disease include progressive muscle weakness and wasting from distal to proximal, ptosis, weakness of facial, jaw and anterior neck muscles, myotonia, daytime sleepiness, fatigue and cataract. Other symptoms of adult DM1 include cardiac conduction defects, as well as endocrine, gastrointestinal and cognitive dysfunction. DM1 is one of the most variable human diseases, has complex, multisystemic and progressively worsening clinical manifestations and leads to severe physical impairment, restricted social participation and premature death.

There is no pharmaceutical treatment for causal or symptomatic relief of DM1 core symptoms (with the exception of Modafinil for excessive daytime sleepiness). Thus the aim of treatment is to relieve impairments, reduce limitations and optimise participation. Physical activity has been acknowledged as an important factor for health in general. For patients with a slowly progressive neuromuscular disease, such as DM1, there is accumulating evidence for prescribing low-to-moderate-intensity strength and aerobic exercise training, and an active lifestyle. Nevertheless, recent reviews conclude that existing studies are limited in number and quality, and that there is a need for disease-specific, randomised, controlled trials investigating the effect on quality of life.

RATIONALE FOR THE STUDY It was demonstrated recently by an OPTIMISTIC research partner that severe fatigue, defined as a score equal to or higher than 35 on the subscale fatigue of the Checklist Individual Strength (CIS-fatigue), was reported by around 70% of patients with DM1. These severely fatigued patients had more problems with physical and social functioning as well as with their mental and general health than similar patients without severe fatigue. They also had more problems with concentration and planning. As such, experienced fatigue should be clearly distinguished from muscle weakness, which is probably the most common and characteristic symptom of DM1 and also of a lack of initiative (apathy) that is known to occur often in DM1.

In a longitudinal study, we built a model of perpetuating factors for fatigue in patients with DM1. It appeared that lack of physical activity, sleep disturbances and pain all contributed to experienced fatigue. In addition, loss of muscle strength and pain contributed to fatigue through a lower level of physical activity. Ultimately, experienced fatigue and physical activity both contributed to the level of societal participation. A lack of initiative further increased fatigue but also had a direct negative effect on societal participation. Thus, theoretically, in order to improve societal participation one should compensate for a reduced initiative, optimise physical activity and alleviate experienced fatigue. To alleviate fatigue one should address the fatigue maintaining factors identified by the model, e.g. experience of pain or sleep disorders.

The main rationale for the combination of CBT and physical activity is based on our DM1-specific model. The DM1-specific model shows that physical activity, experienced fatigue and lack of initiative are the main determinants of DM1 health status. OPTIMISTIC is the first model-based clinical trial in DM1. It evaluates the effect, and the maintenance of effects, of CBT combined with exercise training on the reduction of chronic fatigue in patients with DM1.

Importantly, the intervention will also involve caregivers where they are willing to take part. The disabilities associated with DM1 put considerable strain on caregivers and can also lead to a negative interaction with the patient. The intervention will aim to support caregivers by installing realistic expectations about what can be expected from the patient, teach caregivers how to help patients to stay as self-reliant as possible and also reduce caregivers strain by taking time for themselves. If a DM1 patient has no caregiver or significant other, or no caregiver or significant other willing to take part in the study, the patient will not be excluded from the study. All patients will be asked if the study team could approach them to inform them for further research. This contact does not constitute consent.

** CMRI-substudy in People with DM1 People with DM1 are at high risk of developing a cardiac complication. However, it is not known whether the high prevalence of cardiac complications can be affected by a sedentary lifestyle. Given the high risk of cardiac complications and the possibility that becoming more physically active may help these complications, the University of Newcastle, will conduct a sub-study to perform Cardiac Magnetic Resonance Imaging (CMRI) in 40 eligible participants at baseline and at end of the intervention period to acquire the evidence upon which clinical judgement about the use of exercise as a clinical therapy that is safe, can be based.

Cardiac Magnetic resonance imaging (CMRI) uses a combination of harmless radiofrequency (RF) waves and powerful magnets to cause hydrogen nuclei within the cardiac cell molecules to vibrate and emit RF energy. The MRI scanner detects the energy emissions and converts them to viewable images. When diseases begin, there are changes in the heart's tissue. Because even minor changes in tissue affect the rates at which energy is emitted, many medical conditions can be detected at their very early stages. MRI is done to evaluate the structure and function of the heart and blood vessels. MRI may provide information that cannot be obtained by other tests such as chest X-ray, ECG, echocardiogram, or nuclear tests.

The CMRI examinations will be performed with the contract enhancement gadolinium, in 40 eligible participants, 20 in each group. Participants will undergo:

1. cardiac cine imaging, to evaluate cardiac morphology
2. systolic and diastolic function and
3. cardiac tagging to evaluate wall motion and torsion.

MRI safety will be established prior to baseline and end of intervention scan. This includes; assessing for in vivo ferrous material, claustrophobia, abnormal renal function and pregnancy. The PI will assess renal function from the participant's medical notes at screening, if required a blood tests for U&Es will be requested. In addition, child-bearing potential female participants will consent to have urine pregnancy test performed.

For participants that have had a baseline CMRI and withdraw from the study prior to the end of the intervention period, will be invited to have an end of study CMRI if the period from their initial CMRI is greater than 3 months.

No further statistical review is required for the CMRI sub-study as only frequencies and associations will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Genetically proven DM1
* Suffering from severe fatigue (CIS fatigue >35
* Able to walk independently

Exclusion Criteria:

* Neurological or orthopaedic co-morbidity interfering with the interventions or possibly influencing outcomes.
* Use of psychotropic drugs (except Modafinil, Ritalin and antidepressants where the dosing regimen has been stable for at least 12 months prior to screening). If the doses of Modafinil or Ritalin increase during the 10 months of the intervention then the participant will be excluded.
* Severe depression as screening (judged as meeting DSM-IV criteria for a depressive episode).
* Participation in another clinical trial of an investigational medicinal product (CTIMP) or other interventional study considered to influence outcomes being evaluated in OPTIMISTIC.
* Unable to complete study questionnaires.
* Subject participating in another clinical trial (other than observational trials and registries) concurrently or within 30 days prior to screening for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2016-03-29 (Actual); Study Completion 2016-10-17 (Actual)

PRIMARY OUTCOMES:
DM1-Activ | Baseline and 10 months
  The primary outcome measure will be the change in DM1-Activ score. DM1-Activ is a specific outcome measure of activity and participation for patients with DM1.

SECONDARY OUTCOMES:
Six Minute Walk Test | Baseline and 10 months
  Six minute walk test with BORG scale assessment
Myotonic Dystrophy Health Index (MDHI) | Baseline and 10 months
Physical activity measured with actometer | Baseline and 10 months
Fatigue and Daytime Sleepiness Scale (FDSS) | Baseline and 10 months
Checklist Individual Strength (CIS) | Baseline and 10 months
Individualised Neuromuscular Quality of Life Questionnaire (InQoL) | Baseline and 10 months
Beck depression Inventory for Primary Care | Baseline and 10 months
Apathy Evaluation Scale (AES) | Baseline and 10 months
Stroop Test | Baseline and 10 months

OTHER OUTCOMES:
Explanatory and/or Predictive outcomes | Baseline, 10 and 16 months
  Biomarkers (urine and blood)

CONTACTS AND LOCATIONS:
Overall Officials: Grainne Gorman, Dr, Principal Investigator — Newcastle University; Baziel van Engelen, Prof, Principal Investigator — Radboud University Nijmegen Medical Centre, The Netherlands; Benedikt Schoser, Prof, Principal Investigator — Munich University, Germany; Guillaume Bassez, Prof, Principal Investigator — Assistance Publique-Hospitaux de Paris, France
Locations (4):
- Assistance Publique-Hospitaux de Paris, Paris, France
- Friedrich Naur Institute, Munich, Germany
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands
- Newcastle University, Newcastle, United Kingdom

REFERENCES:
- [Background] van Engelen B; OPTIMISTIC Consortium. Cognitive behaviour therapy plus aerobic exercise training to increase activity in patients with myotonic dystrophy type 1 (DM1) compared to usual care (OPTIMISTIC): study protocol for randomised controlled trial. Trials. 2015 May 23;16:224. doi: 10.1186/s13063-015-0737-7. PMID 26002596
- [Derived] Wenninger S, Cumming SA, Gutschmidt K, Okkersen K, Jimenez-Moreno AC, Daidj F, Lochmuller H, Hogarth F, Knoop H, Bassez G, Monckton DG, van Engelen BGM, Schoser B. Associations Between Variant Repeat Interruptions and Clinical Outcomes in Myotonic Dystrophy Type 1. Neurol Genet. 2021 Mar 9;7(2):e572. doi: 10.1212/NXG.0000000000000572. eCollection 2021 Apr. PMID 33884298
- [Derived] Heskamp L, van Nimwegen M, Ploegmakers MJ, Bassez G, Deux JF, Cumming SA, Monckton DG, van Engelen BGM, Heerschap A. Lower extremity muscle pathology in myotonic dystrophy type 1 assessed by quantitative MRI. Neurology. 2019 Jun 11;92(24):e2803-e2814. doi: 10.1212/WNL.0000000000007648. Epub 2019 May 22. PMID 31118244
- [Derived] Okkersen K, Jimenez-Moreno C, Wenninger S, Daidj F, Glennon J, Cumming S, Littleford R, Monckton DG, Lochmuller H, Catt M, Faber CG, Hapca A, Donnan PT, Gorman G, Bassez G, Schoser B, Knoop H, Treweek S, van Engelen BGM; OPTIMISTIC consortium. Cognitive behavioural therapy with optional graded exercise therapy in patients with severe fatigue with myotonic dystrophy type 1: a multicentre, single-blind, randomised trial. Lancet Neurol. 2018 Aug;17(8):671-680. doi: 10.1016/S1474-4422(18)30203-5. Epub 2018 Jun 19. PMID 29934199
- See also: Website providing Trial Information for patients and professionals — http://optimistic-dm.eu/